CLINICAL TRIAL: NCT00993239
Title: A Phase 1, Open-Label, Non-randomized, Dose Escalation Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of TL32711 in Adults With Refractory Solid Tumors or Lymphoma
Brief Title: Dose Escalation Safety Study of TL32711 in Adults With Refractory Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TetraLogic Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TL32711-FIH-007-PTL-F
Record Dates: First submitted 2009-10-08; First posted 2009-10-12 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — birinapant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Birinapant (TL32711) (Experimental)
  Interventions: Drug: Birinapant (TL32711)

INTERVENTIONS:
Drug: Birinapant (TL32711) — 30 minute intravenous (IV) infusion administered once weekly for three consecutive weeks followed by a one week off (Cycle) repeated every 4 weeks as tolerated
  Other Names: NSC 756502

SUMMARY:
A Phase 1 open-label, non-randomized dose escalation study to determine the maximum tolerated dose (MTD) and characterize the safety and tolerability of Birinapant (TL32711).

DETAILED DESCRIPTION:
The purpose of this Phase 1 open-label, non-randomized dose escalation study is to determine the maximum tolerated dose (MTD) and characterize the safety and tolerability of Birinapant (TL32711) when administered as a 30 minute intravenous infusion once weekly for three weeks per repeated 4 week intervals in subjects with refractory solid tumors or lymphoma. Additionally study will assess anti-tumor activity, pharmacokinetics, and exploratory biomarkers as a measurement of pharmacodynamic effects.

ELIGIBILITY:
Key Inclusion Criteria:

* Advanced metastatic or unresectable malignancy that is refractory to currently available standard therapies or no effective therapy exists. The subject's malignancy must be confirmed by prior pathologic study.
* Evaluable disease (measurable or non-measurable) by Response Evaluation Criteria in Solid Tumors (RECIST, Version 1.1) or Revised Response Criteria for Malignant Lymphoma (RRCML) (Cheson 2007).
* Life expectancy greater than 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Adequate renal function, defined as serum creatinine ≤ 1.5 X upper limit of normal (ULN), or calculated creatinine clearance ≥ 60 ml/min.
* Adequate hepatic function, defined as aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 3 X ULN and total bilirubin < 1.5 X ULN.
* Adequate bone marrow function, defined as absolute neutrophil (ANC) ≥ 1,500/mm3 (≥1.5 X106/L), platelet count ≥ 75,000/mm3 (≥ 75 X106/L), and hemoglobin ≥ 10 mg/dL in the absence of transfusion.

Key Exclusion Criteria:

* Recent anti-cancer treatment defined as:

  * Standard or investigational anti-cancer therapy within 4 weeks prior to first dose of TL32711. Exception: continued hormonal interventions for sensitive diseases.
  * Radiation therapy within 2 weeks prior to the first dose of TL32711.
* Clinically significant pulmonary illness resulting in Grade ≥ 2 hypoxia (National Cancer Institute Common Terminology criteria for Adverse Events [NCI CTCAE, v4]) or any requirement for supplemental oxygen, or pulse oximetry less than 90% saturation on room air.
* Symptomatic or uncontrolled brain metastases requiring current treatment (less than 4 weeks from last cranial radiation or 2 weeks from last steroids).
* Impaired cardiac function or clinically significant cardiac disease.
* Ongoing auto-immune disease or with history of an auto-immune disease within the past 5 years. Auto-immune disease include but are not limited to systemic lupus erythematosis, scleroderma, rheumatoid arthritis, psoriasis, psoriatic arthritis, ulcerative colitis and regional enteritis (Crohn's disease).
* Systemic or chronic topical corticosteroids or immunosuppressive therapy within 4 weeks prior to study entry or anticipated need of systemic corticosteroids or immunosuppressive therapy during study participation.
* Skin lesions of Grade ≥ 2 severity (NCI CTCAE v4), except alopecia.
* Lack of recovery of prior adverse events to Grade ≤1 severity (NCI CTCAE v 4) (except alopecia or neuropathy) due to medications administered prior to the first dose of TL32711.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-11; Primary Completion 2012-08 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Define the MTD | 4 weeks (Cycle 1)

SECONDARY OUTCOMES:
Tumor burden according to Response Evaluation Criteria in Solid Tumors (RECIST)/Revised Response Criteria Malignant Lymphoma | Every 8 weeks (2 cycles) while on treatment
Translational biomarkers and pharmacokinetics | First and third dose of Cycle 1 and after every two cycles (biomarkers only) while on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Amaravadi, MD, Principal Investigator — University of Pennsylvania, Abramson Cancer Center; Lainie P Martin, MD, Principal Investigator — Fox Chase Cancer Center; Alex Adjei, MD, PhD, Principal Investigator — Roswell Park Cancer Institute
Locations (3):
- United States (3):
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania